CLINICAL TRIAL: NCT04773210
Title: Association Between Type of Ligating Brackets and Oral Health-related Quality of Life in Orthodontic Patients
Acronym: OHIPS14ORTHO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundación Universitaria CIEO (Other)
Responsible Party: Sponsor
Other Study IDs: UniCIEO OHIP-S14 ORTHO
Record Dates: First submitted 2021-02-23; First posted 2021-02-26 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Oral Health-related Quality of Life; Orthodontic Treatment
Keywords: Health-Related Quality of Life; Oral Health Impact Profile; Orthodontics, Corrective; Orthodontic Appliances

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Mini tube system: Mini tube system (FLOW-JAC System, Bogotá, Colombia) orthodontic treatment.
  Interventions: Device: Mini tube system
- Conventional ligating brackets: Conventional ligating brackets (Gemini 3M Unitek Orthodontic Products bracket, Calif, USA) with Nitinol Classic or superelastic (SE) archwires 0.014 and 0.016 orthodontic treatment.
  Interventions: Device: Conventional ligating brackets

INTERVENTIONS:
Device: Mini tube system — Mini tube system (FLOW-JAC System, Bogotá, Colombia) orthodontic treatment
  Groups: Mini tube system
Device: Conventional ligating brackets — Conventional ligating brackets (Gemini 3M Unitek Orthodontic Products bracket, Calif, USA) with Nitinol Classic or superelastic (SE) archwires 0.014 and 0.016 orthodontic treatment
  Groups: Conventional ligating brackets

SUMMARY:
To evaluate the association of the level of quality of life related to oral health, between treatment with the minitube system and conventional ligation brackets, in adult patients with moderate malocclusion, during the first six months, of orthodontic treatment.

DETAILED DESCRIPTION:
This is an observational cohort study with 1: 1 allocation ratio. The sample will be of 200 participants, divided into two groups. People over 18 years of age will be included; with moderate treatment complexity determined by Dental Aesthetics Index DAI. The study interventions are: (1) Mini tube system (FLOW-JAC System, Bogotá, Colombia) and (2) Conventional ligating brackets (Gemini 3M Unitek Orthodontic Products bracket, Calif, USA) with Nitinol Classic or superelastic (SE) archwires 0.014 and 0.016.

The outcome variable is Oral health-related quality of life (OHRQoL) measured with OHIP-S14 Ortho instrument, which was validated in Spanish in patients with orthodontic treatment. Consists of 14 questions that address seven dimensions (functional limitation, physical pain, psychological discomfort, physical disability, psychological disability, social disability and handicap), specifically related to orthodontic treatment. The OHIP-S14 Ortho score is between 0 to 56. Where 0 indicates a positive impact and 56 an unfavorable impact. The questionnaire will be self-administered online during the first 6 months of treatment: T0: prior to cementation, T1: 24 -48 hours after cementation, T2: 1 month after cementation, T3: 3 months after cementation and T4: 6 months after cementation.

ELIGIBILITY:
Inclusion Criteria:

* Age range from 18 to 35
* Moderate treatment complexity determined by Dental Aesthetics Index DAI moderate.
* Orthodontic treatment with mini tube system in upper and lower jaw or MBT conventional ligating pre-set appliances
* Non- extractions at the start of orthodontic treatment
* Non- placement of mini-implants at the start of orthodontic treatment

Exclusion Criteria:

* Craniofacial anomalies
* Dental caries at the start of orthodontic treatment
* Periodontal disease at the start of orthodontic treatment
* Systemic disease
* Orthognathic surgery indicated
* Cognitive disorders
* Non understand the Spanish language

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients wearing orthodontic treatment with mini tube system in upper and lower jaw or MBT conventional ligating pre-set appliances
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-04-12 (Actual); Primary Completion 2022-11-19 (Estimated); Study Completion 2023-02-18 (Estimated)

PRIMARY OUTCOMES:
Oral health-related quality of life (OHRQoL) | Change from baseline to 6 months
  Oral health-related quality of life (OHRQoL) measured with OHIP-S14 Ortho instrument, which was validated in Spanish in patients with orthodontic treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Plaza, MSD, Principal Investigator — Fundación Universitaria CIEO
Locations (1):
- Fundación Universitaria CIEO Uni-CIEO, Bogotá, Colombia

IPD SHARING:
Plan to Share IPD: No